CLINICAL TRIAL: NCT03059134
Title: Therapeutic Efficacy and Safety of Mirabegron , a β3-Adrenoceptor Agonist, Treatment on Patients With Overactive Bladder Syndrome in Taiwan - Predictive Factors for the First Line Use and the Dose Effectiveness Relationship
Brief Title: Mirabegron Treatment on Patients With Overactive Bladder Syndrome in Taiwan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Hann-Chorng Kuo, Chairman, Department of Urology, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BuddhistTCGH
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Urinary Incontinence; Overactive Bladder Syndrome
Keywords: Overactive bladder; Pharmacotherapy; Adverse event
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive | interventions — mirabegron

STUDY DESIGN:
Intervention Model Description: The study population consisted of male and female outpatients meeting the legal minimum age requirement of the region with symptoms of OAB for more than 3 months. Patient demographics data will be recorded as detailed as possible, including previous urodynamic study results. The study consisted of four arms:
  1. Mirabegron 25mg once-daily for 4 weeks, and continue the same dose of mirabegron for another 8 weeks
  2. Mirabegron 25mg once-daily for 4 weeks, and increase the dose to 50mg for another 8 weeks
  3. Mirabegron 25mg once-daily for 4 weeks, and shift to solifenacin 5mg for another 8 weeks
  4. Mirabegron 25mg once-daily for 4 weeks, and add-on solifenacin 5mg for another 8 weeks,
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Mirabegron 25mg for 12 weeks (Experimental): Mirabegron 25mg once-daily for 4 weeks, and continue the same dose of mirabegron for another 8 weeks
  Interventions: Drug: Mirabegron 25mg
- Mirabegron 25mg followed by 50mg (Active Comparator): Mirabegron 25mg once-daily for 4 weeks, and increase the dose to 50mg for another 8 weeks
  Interventions: Drug: Mirabegron 25mg
- Mirabegron 25mg followed by solifenacin (Active Comparator): Mirabegron 25mg once-daily for 4 weeks, and shift to solifenacin 5mg for another 8 weeks
  Interventions: Drug: Mirabegron 25mg
- Mirabegron 25mg add-on solifenacin (Active Comparator): Mirabegron 25mg once-daily for 4 weeks, and add-on solifenacin 5mg for another 8 weeks,
  Interventions: Drug: Mirabegron 25mg

INTERVENTIONS:
Drug: Mirabegron 25mg — We compared the therapeutic effects and adverse events (AEs) in overactive bladder (OAB) patients receiving different combination of mirabegron and solifenacin.
  Other Names: Betmiga

SUMMARY:
This clinical trial compared the therapeutic effects and adverse events (AEs) in overactive bladder (OAB) patients receiving different combination of mirabegron and antimuscarinics.

Methods: This is a prospective randomized study. OAB patients received mirabegron 25 mg (M25) daily for one month (1M) and then were randomized as group 1: to continue M25, group 2: to mirabegron 50 mg, group 3: to shift to solifenacin 5 mg (S5) and group 4: to combine M25 and S5 for further 2 months (totally 3 months, 3M). Efficacy and AEs were evaluated. At the end of 3M, the preferred option for future treatment was investigated.

DETAILED DESCRIPTION:
Introduction

Overactive bladder syndrome (OAB) is defined as the symptom syndrome with frequency, and urgency with or without urgency incontinence. OAB affects more than 400 million people worldwide and has been estimated to affect around 16% of the adult population across Europe and the USA. In Asian countries, the prevalence of OAB has been reported to be 6% of men and women aged ≥18 years in China; 12.2% of men and women in Korea;12.4% of men and women aged ≥40 years in Japan; and 21 to 25% of women and 16.9% of community dwelling adults in Taiwan. Another study reported that the prevalence of OAB among adult men across 11 Asian countries (India, Indonesia, Malaysia, Pakistan, Philippines, Singapore, South Korea, Taiwan, China, Hong Kong and Thailand) was 29.9%.

Antimuscarinics are first line pharmacotherapy for OAB. However, some patients have a suboptimal response to antimuscarinics and some may experience adverse effects, such as dry mouth or constipation. Therefore, a high proportion of patients discontinue antimuscarinic therapy, with fewer than 25% remaining on treatment at 1 year. There is an unmet need to develop new drugs for OAB without the bothersome adverse effects of antimuscarinic agents.

β3-adrenergic receptors are known to promote urine storage in the bladder by inducing detrusor relaxation in animal and human bladders. In humans, the β3-adrenoceptor is the predominant β-receptor subtype in the urinary bladder. β3-adrenoceptor agonists relax the detrusor smooth muscle during the bladder storage phase and increase bladder capacity without accompanying changes in micturition pressure, residual volume or voiding contraction.

Mirabegron is the first β3-adrenoceptor agonist to have been approved for the treatment of OAB. Pooled safety data indicates that dry mouth, the chief cause of treatment discontinuation with antimuscarinic agents, occurs with low incidence with mirabegronc. Hence, mirabegron may be a valuable treatment option for patients with OAB.

Recent phase III trials have confirmed the efficacy and safety of mirabegron in the treatment of OAB in Europeans, Australians, North Americans, Japanese and Asians. Whether mirabegron should be used as the first line treatment for OAB has not been determined yet. There is also no study showing that mirabegron is superior to solifenacin in terms of therapeutic efficacy and safety profile. The dose effectiveness relationship between 25mg and 50mg mirabegron has also not been investigated yet. Hence, we have conducted this post marketing study in order to evaluate the efficacy and safety of mirabegron in Taiwanese people with symptoms of OAB.

Materials and Methods

Study design and participants

This prospective, randomized trial will be conducted in Tzu Chi General Hospital, Hualien, Taiwan. The study population consisted of male and female outpatients meeting the legal minimum age requirement of the region with symptoms of OAB for more than 3 months. Patient demographics data will be recorded as detailed as possible, including previous urodynamic study results.

The study consisted of four arms:

1. Mirabegron 25mg once-daily for 4 weeks, and continue the same dose of mirabegron for another 8 weeks
2. Mirabegron 25mg once-daily for 4 weeks, and increase the dose to 50mg for another 8 weeks
3. Mirabegron 25mg once-daily for 4 weeks, and shift to solifenacin 5mg for another 8 weeks
4. Mirabegron 25mg once-daily for 4 weeks, and add-on solifenacin 5mg for another 8 weeks,

Randomization was accomplished using a computer-generated randomization scheme (Cenduit GmbH, Allshwil, Switzerland) with stratification by site; allocation to treatment groups at each site was accomplished via an interactive response system with a study coordinator. Study visits took place at Week 0 (Visit 1; confirmation of eligibility criteria); Weeks 4, 8 and 12 (Visits 2, 3 and 4).

The study was approved by the institutional review board of each study site and conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki, Good Clinical Practice, International Conference on Harmonisation guidelines, and all applicable laws and regulations.

The sample size for this study was based on results from a 12-week dose-finding Phase II study (178-CL-045; NCT00527033) conducted in Japan. In that study, the mean decrease of urgency episodes per 24 hours for the mirabegron 50mg group was 2.24. The primary efficacy end-point in this study is the percentage of patients with a change from baseline to the final visit in the urgency episodes per 24 hours by 2 or greater. The number of patients per group necessary to demonstrate superiority to the first group (mirabegron 25mg for 12 weeks) would be 263 with an effect size of 0.2, at a two-sided significance level of 5% and power of 90%. Assuming a dropout rate of 15% during the treatment period, 302 subjects per group are to be enrolled for randomization.

The results of this study will provide evidence for the sup[eriority of which medicatyion and combination of pharmacotherapy in treatment of patients with overactive bladder syndrome. We also expected to search for the predictive factors for responders to mirabegron 25mg alone, mirabegron 50mg, solifenacin alone, and combined mirabegron 25mg an slifenacin 5mg, based on the baseline demographics and urodynamic study findings

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms of OAB for at least 12 weeks before initiation of the run-in period;
2. An average of ≥8 micturitions per 24 hours,
3. An average of ≥1 episode of urgency or urgency incontinence per 24-hours, during a 3-day micturition diary period.

Exclusion Criteria:

1. Stress urinary incontinence as a predominant symptom at screening;
2. Urinary tract infection, urinary stone, interstitial cystitis or a history of recurrent urinary tract infection;
3. Confirmed post-void residual (PVR) volume of ≥100 mL or more or with a clinically significant lower urinary tract obstructive disease;
4. Proven neurogenic bladder such as stroke, Parkinson's disease, spinal cord injury, multiple sclerosis;
5. Overt bladder outlet obstruction not adequately controlled.
6. Severe medical disease that prohibit patients to undergo clinical investigation.
7. Patient is currently taking medications that might affect lower urinary tract function, such as α1-adrenoreceptor antagonists; medication for diabetes insipidus, antidepressants, 5α reductase inhibitors, capsaicin, resiniferatoxin, or botulinum toxin into the bladder, were also restricted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2016-04-27 (Actual); Study Completion 2016-04-27 (Actual)

PRIMARY OUTCOMES:
Reduction of urgency or urgency incontinence episode by 2 per day | from baseline to 12 weeks
  The percentage of patients in each arm who had reduction of urgency or urgency incontinence episode by 2 per day

SECONDARY OUTCOMES:
International Prostate Symptom Score total (IPSS-T) | from baseline to 12 weeks
  The change of the general bladder symptom score
quality of life (QoL) index | from baseline to 12 weeks
  The change of QoL index
Overactive Bladder Symptom Score (OABSS) | from baseline to 12 weeks
  The change of OABSS
Urgency Severity Scale (USS) | from baseline to 12 weeks
  The change of USS
Patient's Perception of Bladder Condition (PPBC) | from baseline to 12 weeks
  The change of PPBC
Global Response Assessment (GRA) | from baseline to 12 weeks
  The change of GRA
maximum flow rate (Qmax) | from baseline to 12 weeks
  The change of Qmax
voided volume (Vol) | from baseline to 12 weeks
  The change of vol
Postvoid residual volume m(PVR) | from baseline to 12 weeks
  The change of PVR

CONTACTS AND LOCATIONS:
Overall Officials: Hann-Chorng Kuo, MD, Principal Investigator — Department of Urology, Buddhist Tzu Chi General Hospital, Hualien, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD was not planned to share